CLINICAL TRIAL: NCT01540019
Title: Guarana (Paullinia Cupana) for Anorexia Related to Cancer
Brief Title: Paullinia Cupana for Anorexia in Oncologic Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Felipe Melo Cruz, MsC, Faculdade de Medicina do ABC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FaculdadeMABC
Record Dates: First submitted 2012-01-29; First posted 2012-02-28 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-01

CONDITIONS: Cancer-related Problem/Condition; Anorexia; Loss of Weight
Keywords: anorexia; Paullinia cupana; loss of weight
MeSH Terms: conditions — Anorexia; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paullinea cupana (Experimental): 50mg of Paullinia cupana as capsule, twice daily
  Interventions: Drug: Paullinia cupana

INTERVENTIONS:
Drug: Paullinia cupana — 50mg of Paullinia cupana as capsule, twice daily

SUMMARY:
Denutrition, lost of weight and anorexia are present in many oncologic patients at any time of the disease. Anorexia is the spontaneous loss of appetite and many changes in the metabolism are made in this case, leading to this syndrome called anorexia-cachexia, that includes changes in the tumoral response and inflammatory pathways. The guaraná (Paullinia cupana) is originally from Brazil and Venezuela and has been used culturally for headaches, muscle pains, depression and others. As it has shown a good response and tolerability for fatigue, the investigators decide to try guaraná for anorexia. Patients will receive guaraná as capsules of 50 mg twice daily, for 4 weeks, and will be weighted and respond questionaries about quality of life.

DETAILED DESCRIPTION:
Patients 18 years and older, diagnosed with any cancer, that is losing weight and have anorexia will be selected. They must have normal levels of creatinine, thyroid evaluation and hepatic function. If they are taking corticosteroid, they must keep losing weight and refer anorexia, as well as if they are on treatment with chemotherapy.

Patients will receive 50mg of the guaraná twice daily for 4 weeks. Every week will be an evaluation of the weight, level of appetite and answer 2 questionaries of quality of life and level of symptoms (FACT-G and MDASI).

This is a fase II study, open-label, no randomized, with two steps following ¨two stages of Simon¨ model. First step 18 patients will be included and if there are 3 good responses second step will follow, including 17 more patients. Response will be considered if there is at least 5% of gain in the weight.

ELIGIBILITY:
Inclusion Criteria:

* adults (18 years old and older)
* palliative care or oncologic treatment
* loss of weight
* anorexia

Exclusion Criteria:

* gastrointestinal obstruction
* blood pressure not controlled
* diabetes not treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
weight | eight weeks
  Patients will considered to respond to guaraná if the gain 5% or more of his inicial weight during the treatment period

SECONDARY OUTCOMES:
quality of life | eight weeks
  Weekly patients will answer questionaries about quality of life like FACT-G

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Latorre, Study Chair — Faculdade de Medicina do ABC
Locations (1):
- Faculdade de Medicina do ABC, Santo André, São Paulo, Brazil